CLINICAL TRIAL: NCT04958876
Title: Phase 1, Double-blind, Randomized, 2-Period, 2-Treatment Crossover Study to Evaluate the Safety of SP-104 Compared to Immediate Release Naltrexone Capsules in Healthy Adult Subjects
Brief Title: Study to Evaluate the Safety of SP-104
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scilex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP-104-02
Record Dates: First submitted 2021-07-06; First posted 2021-07-12 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Dronabinol; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SP-104 crossover to naltrexone immediate release (Experimental): SP-104 administration followed by a crossover to naltrexone immediate release oral capsule administration
  Interventions: Drug: SP-104; Drug: Naltrexone immediate release oral capsules
- Naltrexone immediate release crossover to SP-104 (Experimental): Naltrexone immediate release oral capsule administration with a crossover to SP-104 administration
  Interventions: Drug: SP-104; Drug: Naltrexone immediate release oral capsules

INTERVENTIONS:
Drug: SP-104 — oral capsule once daily
Drug: Naltrexone immediate release oral capsules — oral capsule once daily

SUMMARY:
Evaluate the safety and tolerability of 3-day repeat-dose of SP-104 compared to naltrexone hydrochloride immediate release.

DETAILED DESCRIPTION:
The purpose of this trial is to evaluate the safety and tolerability of SP-104 relative to naltrexone immediate release capsules in healthy adults. The study is designed to test the hypothesis that the formulation of SP-104 will mitigate against adverse events associated with naltrexone.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to read, write, and understand the English language and provide English language written informed consent (IC) prior to beginning any study procedures.
2. Male or female age 18 to 70 years (inclusive) at screening.
3. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or electrocardiogram (ECG), as deemed by the Investigator.
4. Negative urine drug screen for drugs of abuse, including cocaine, marijuana, amphetamines, and barbiturates at the Screening Visit and at each check-in.
5. If female, heterosexually active, of childbearing potential, not pregnant, not trying to become pregnant, or lactating, individuals are eligible to participate if participants agree to total abstinence from heterosexual intercourse, from screening through until at least 30 days after the last study dose, or to the use of an effective method listed below, from screening through until at least 30 days after the last study dose. A second non-hormonal method of contraception is required if a hormonal form of birth control is used. Females of childbearing potential must have negative pregnancy tests at Screening and on admission.
6. If male and heterosexually active, individuals are eligible to participate if participants agree to total abstinence from heterosexual intercourse, from screening through until at least 90 days after the last study dose, or to the use of an effective method listed below, from screening through until at least 90 days after the last study dose.
7. Able to swallow capsules.
8. Agrees to comply with all study requirements throughout the entire study period.

Exclusion Criteria:

1. A body mass index (BMI) <18 kg/m2 or >30 kg/m2 (without rounding).
2. Are using prescription medications or over-the-counter products (including dietary supplements such as vitamins, minerals, herbs or other botanicals, amino acids, enzymes (extracts or concentrates), or probiotics (bacteria or yeasts), within 14 days prior to administration of the study medication.
3. Currently using or have recently used opioids
4. Use of any other investigational drug within 30 days prior to administration of the study medication.
5. History of allergic or adverse response to naltrexone.
6. History of drug or alcohol abuse (>80 g/day).
7. History of sleep apnea or restless leg syndrome.
8. Serology positive for hepatitis B surface antigen, hepatitis C antibodies, or human immunodeficiency virus (HIV) antibodies.
9. Positive for known disease (e.g., corona virus disease 2019 (COVID-19 )).
10. Subjects with current or past SARS-CoV-2 infection, if tested according to local requirements.
11. Have had a serious illness in the 4 weeks preceding the Screening Visit that resulted in missed work or hospitalization (note: missed work in itself may not denote serious illness).
12. Have cancer within the past 5 years (treated or untreated).
13. Are females who are pregnant, plan to become pregnant during the study, or are breastfeeding.
14. Are an employee, family member, sponsor, or student of the Investigator or of the clinical site.
15. Are unable to understand or adhere to the requirements of the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | 1 week

CONTACTS AND LOCATIONS:
Locations (2):
- New Zealand (2):
  - Auckland Clinical Studies (NZCR), Auckland
  - Christchurch Clinical Studies Trust (NZCR), Christchurch

IPD SHARING:
Plan to Share IPD: No